CLINICAL TRIAL: NCT00596700
Title: Capsule Endoscopy Crohn's Disease Activity Index - Validation Multi Center Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Rambam Health Care Campus (Other); Assaf-Harofeh Medical Center (Other Government); Hillel Yaffe Medical Center (Other Government); University of Athens (Other); University of Magdeburg (Other)
Responsible Party: Principal Investigator, Yaron Niv, Director Department of Gastroenterology, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CECDAI-2006
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Crohn's Disease
Keywords: Capsule endoscopy; Crohn's disease; IBD; Activity score; Small bowel; Crohn's disease of the small bowel in any stage; Recruiting
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device (Experimental): Patient preparation procedure will be done according to chapter 4 in the Given Diagnostic System user manual. In brief: to drink only clear liquids beginning 12:00 noon the day before.at least 8 hours (since 12:00 PM) fast prior to the procedure. Patient will undergo a standard capsule endoscopy. Patients will be allowed to drink clear liquids 2 hours post ingestion, and eat 4 hours post ingestion.
  Eight hours post ingestion, data recorder will be removed and the patient will be dismissed.
  A local experienced reader will review the RAPID video to determine the diagnosis blinded to the results of the standard workup procedures, and to each other results. Results will be recorded in the case report forms. A decoded video will be transferred to the principal investigator for reevaluation
  Interventions: Device: Given® Diagnostic System including PillCamTM SB Capsules

INTERVENTIONS:
Device: Given® Diagnostic System including PillCamTM SB Capsules — Device for detection of pathologies as a tool in the diagnosis of gastrointestinal disorders.
  An ingestible,disposable video camera that transmits high quality images of the small intestinal mucosa
  Other Names: PillCam™SB capsule (Given Imaging Ltd, Yoqneam, Israel)

SUMMARY:
The Study

1. Prospective trial of the Niv score validating score against known activity indices - see addendum A for Niv score
2. Known Crohn's disease patients undergoing capsule endoscopy are identified - see addendum B for inclusion/exclusion criteria
3. Prior to capsule exam, temperature is taken, height and weight measured, bloods are drawn for albumin, ESR, HCT, CRP
4. Prior to capsule exam, symptom/exam questionnaire is completed - see addendum C for questionnaire
5. Capsule exam is performed
6. CD of de-identified is made at the study site.
7. Landmarks are confirmed and the small bowel transit time is divided into 2 and labeled on thumbnails
8. CDs are copied
9. CDs of study patients are provided to blinded readers

DETAILED DESCRIPTION:
The Niv score was devised to measure mucosal disease activity in Crohn's disease using capsule endoscopy. This scoring index is based on inflammatory score parameters: Erythema, hyperemia, edema, denudation, nodularity, apthae, erosion, ulcer, bleeding), extent score: Focal, patchy, diffuse, and stricture score: single-passed, multiple-passed, obstruction. The higher the score, the more involvement is observed. The advantage of this index is that it actually measures disease activity and not symptoms in an easy non-invasive manner. For assessing Crohn's disease, mucosal healing can be directly seen and if there is no mucosal disease there can be no symptoms secondary to inflammatory bowel disease. The subjective nature of disease activity indices is avoided, as is the problem of disease without symptoms. It is envisioned that the Niv score could diagnose Crohn's disease (excluding normally occurring mucosal breaks), identify NSAID damage, measure disease activity / severity, measure drug response for clinical trials and in practice, and guide medical management for the patient's with small bowel Crohn's disease.

This study will measure the Niv score against CDAI. Since capsule endoscopy assesses mucosal disease and not symptoms it is not envisioned that the Niv score will perfectly correlate with the Harvey-Bradshaw score. It is envisioned that the Niv score will have the same direction. Both of these indices will be determined as part of a multicenter trial. The trial design is outlined below.

The Study

1. Prospective trial of the Niv score validating score against known activity indices - see addendum A for Niv score
2. Known Crohn's disease patients undergoing capsule endoscopy are identified - see addendum B for inclusion/exclusion criteria
3. Prior to capsule exam, temperature is taken, height and weight measured, bloods are drawn for albumin, ESR, HCT, CRP
4. Prior to capsule exam, symptom/exam questionnaire is completed - see addendum C for questionnaire
5. Capsule exam is performed
6. CD of de-identified is made at the study site.
7. Landmarks are confirmed and the small bowel transit time is divided into 2 and labeled on thumbnails
8. CDs are copied
9. CDs of study patients are provided to blinded readers

   Scoring sheets will be provided to readers - see addendum A
10. Readers will score the CDs and return the scoring sheets to the principal investigator
11. Data is collated and analyzed

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older and not greater than 80 years suffer from Crohn's Disease of the small bowel, documented by clinical, endoscopical, histopathological and radiological parameters, in any activity stage iof the disease and any treatment
* Documented written Informed Consent

Exclusion Criteria:

* Subject suffers from swallowing difficulties
* Female subject is pregnant or nursing (in case of necessary small bowel series a pregnancy test has to be performed prior to the test)
* Subject is known to suffer from intestinal obstruction
* Subject has a cardiac pacemakers or other implanted electro medical devices
* Patients with more than 40% small bowel resect
* Subject has any condition, which precludes compliance with study and/or device instructions
* Subject suffers from life threatening conditions
* Subject is currently participating in another clinical study
* Subject with colonic involvement of Crohn's disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
This prospective study is aimed to evaluate the correlation of capsule endoscopy CECDAI with the CDAI (accepted clinical index) and IBDQ (quality of life questionnaire) in patients suffering from small-bowel Crohn's disease | Two years

SECONDARY OUTCOMES:
Capsule endoscopy investigation and crohn's disease outcome | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Niv, MD, AGAF, Principal Investigator — RMC, Tel Aviv University
Locations (4):
- Triniti College, Dublin, Ireland
- Israel (3):
  - Hillel Jafa Medical Center, Hadera
  - Rabin Medical Center, Beilinson Hospital, Tel Aviv University, Petah Tikva
  - Asaf Harofe Medical Center, Zrifin